CLINICAL TRIAL: NCT00927212
Title: Randomized Double Blind Uncontrolled Pilot Study to Compare 2% and 4% AS101 Ointment for the Treatment of Atopic Dermatitis
Brief Title: Topical Application of AS101 for the Treatment of Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial started and halted due sponsor's considerations.
Sponsor: BioMAS Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #76 REV 00
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2011-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 2% AS101 ointment
  Interventions: Drug: AS101 ointment
- Group 2 (Experimental): 4% AS101 ointment
  Interventions: Drug: AS101 ointment

INTERVENTIONS:
Drug: AS101 ointment — Twice daily topical application

SUMMARY:
Atopic Dermatitis is a chronic non contagious disease that causes itchy, inflamed skin. The purpose of this study is to evaluate the safety and efficacy of topical AS101 ointment for the treatment of Atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is the most common chronic inflammatory skin disease, affecting 10-20% of children and 2% of adults worldwide. The mechanism of AD is still not completely understood, but the disorder appears to result from the complex interaction between immunological responses, various susceptability genes, defects in skin barrier function, host and environmental factors and infectious agents. AS101 is a non toxic potent immunomodulator that has been shown to have beneficial effects in diverse pre clinical and clinical studies. Recently, AS101 has shown efficacy and safety in the treatment of mild to moderate Psoriasis which shares with AD a related immunological mechanism along with the AS101 ability to decrease the level of interleukins known to be involved ith the pathogenesis of AD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Atopic Dermatitis for at least 6 months prior to enrollment.
* Diseased Body surface area (BSA) ≤ 20%.
* Male and Female ≥ 18.
* Adequate general health.
* Signed Informed consent form by the patient or his/her legal guardian.
* Patient must be able and willing to comply with all protocol requirements.

Exclusion Criteria:

* Patient who is unable to provide fully informed consent.
* Pregnant of breast-feeding females.
* Concomitant dermatologic or medical condition(s) which may interfere with the patient's response evaluation.
* Evidence of an infection in the targeted zones.
* Known sensitivity to any of the drug component.
* Immunocompromised patients.
* Concomitant medications such as:

  * Topical corticosteroid within 2 weeks prior to Day 1 visit;
  * Systemic steroids and immunosuppressants within 1 month prior to Day 1 visit; *Systemic anti-histamines and antibiotics within 2 weeks prior to Day 1 visit; *Phototherapy within 4 weeks prior to Day 1 visit;
  * Anticipated exaggerated exposure to sunlight during the whole treatment period and 4 weeks prior to Day 1 visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Modified SCORAD index | within 6 weeks treatment and 4 weeks follow up

SECONDARY OUTCOMES:
Remission period | within 4 weeks post treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Felix Pavlotsky, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Dermatology department, Sheba Medical Center, Ramat Gan, Israel